CLINICAL TRIAL: NCT03646071
Title: A Phase 1, Open-label Study of the Safety, Pharmacokinetics and Efficacy of RX108 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of RX108 in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP-102
Record Dates: First submitted 2018-07-18; First posted 2018-08-24 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Locally Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: Locally Advanced; Metastatic; Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Experimental): The Dose-Escalation Phase will employ a standard 3+3 algorithm to investigate ascending dose cohorts of RX108.
  Interventions: Drug: RX108
- Dose Expansion Phase (Experimental): In the Expansion Phase, subjects will receive RX108 at the maximum tolerated dose.
  Interventions: Drug: RX108

INTERVENTIONS:
Drug: RX108 — RX108

SUMMARY:
RX108 is a novel, potent, small-molecule inhibitor of Na+/K+-ATPase. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and efficacy of RX108 in patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a open-label, two-part study comprised of a dose escalation part and a dose expansion part. In the dose escalation part, RX108 will be administered in ascending doses to evaluate the safety and tolerability of RX108 and determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D). The dose expansion part will assess the safety, pharmacokinetics, and efficacy of RX108 at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic cancer that has failed all systemic therapies known to confer clinical benefit
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Minimum age of 18 years
* Adequate hematologic, hepatic and renal function
* Written Informed Consent
* Must agree to use adequate contraception (females and males)

Exclusion Criteria:

* History of certain cardiac abnormalities
* History of inadequate pulmonary function
* Symptomatic brain metastasis
* Treatment with prohibited medications
* Known contra-indication to digoxin
* Treatment with any unapproved therapies for cancer, or any other anti-cancer therapy within 3 weeks
* Any toxicity related to prior treatment must have resolved to Grade 1 or less, with the exception of alopecia
* Clinically significant active infection requiring systemic antibiotic treatment
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum tolerated dose (MTD) of RX108 | Day 1 to 30
  All patients treated with RX108 across all dosing levels will have safety assessed in order to determine the MTD.
Part 2: Incidence of adverse events (AEs) and serious adverse events (SAEs). | Day 1 to 30 days post last dose
  The incidence of adverse events (AEs) and serious adverse events (SAEs) for each cohort dose will be assessed using CTCAE v 5.0.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of RX108 | Day 1 and Day 3: Hours 0, 1, 2, 3, 5, 8
  Pharmacokinetics parameter
Time to reach maximum concentration (Tmax) | Day 1 and Day 3: Hours 0, 1, 2, 3, 5, 8
  Pharmacokinetics parameter
Area under the plasma concentration-time curve (AUC) | Day 1 and Day 3: Hours 0, 1, 2, 3, 5, 8
  Pharmacokinetics parameter
Elimination half-life (T1/2) | Day 1 and Day 3: Hours 0, 1, 2, 3, 5, 8
  Pharmacokinetics parameter
Systemic clearance (CL) | Day 1 and Day 3: Hours 0, 1, 2, 3, 5, 8
  Pharmacokinetics parameter
Response rate (per RECIST v1.1) | Screening and every 2 cycles for the first 6 cycles and every 3 cycles thereafter (each cycle is 28 days), assessed up to 24 months.
  Evaluate the preliminary efficacy of RX108 in subjects with locally advanced or metastatic solid tumors (subjects with measurable disease in Part 2).

CONTACTS AND LOCATIONS:
Overall Officials: Lyon Gleich, MD, Study Director — Medpace, Inc.
Locations (2):
- United States (2):
  - Cedars-Sinai, Los Angeles, California
  - University of Texas at MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
To be determined.